CLINICAL TRIAL: NCT06311422
Title: A 3-Year Clinical Evaluation Of Endocrown Restorations With Two Different Materials Using The Computer-Aided Design/ Computer-Aided Manufacture (Cad/Cam) System
Brief Title: A 3-Year Clinical Evaluation Of Endocrown Restorations With Two Different Materials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Simge Canatan, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAD/CAM-endocrown
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Endodontically Treated Teeth
Keywords: CAD/CAM; Endocrown; resin nanoceramic; zirconia-reinforced lithium silicate
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lava Ultimate block (Experimental): Resin nanoceramic block
  Interventions: Other: resin nanoceramic block
- Celtra Duo block (Active Comparator): zirconia-reinforced lithium silicate block
  Interventions: Other: zirconia-reinforced lithium silicate

INTERVENTIONS:
Other: resin nanoceramic block — Resin-based CAD/CAM materials
  Other Names: Lava Ultimate block
  Arms: Lava Ultimate block
Other: zirconia-reinforced lithium silicate — zirconia reinforced lithium silicate ceramic
  Other Names: Celtra Duo block
  Arms: Celtra Duo block

SUMMARY:
The clinical performance of two different materials in endodontically treated teeth produced with CAD/CAM system will be evaluated and compared. After obtaining a signed informed consert form from all the patients, all restorations will be placed by a single clinician. All endocrown restorations will be produced using the same CAD/CAM system. 52 restorations will be fabricated using Lava Ultimate (LU, 3M Espe, Seefeld, Germany) blocks and 38 restorations will be fabricated using Celtra Duo (CD, Dentsply Sirona, York, PA, USA) blocks. All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using modified United States Public Health Service (USPHS) criteria after baseline, 6,12,36, 48, 60 months. Descriptive statistics will be performed using Chi-square and Fisher exact test.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Patients older than 18
* Teeth must receive endodontic therapy before restoration
* The periodontal condition had to be stabilized before restoration
* No subject complained of discomfort in teeth
* Radiograph revealing alveolar bone resorption of less than a third and no shadow around the periapical tissues
* Participants who provided writen informed consent were recruited in collaboration

Exclusion Criteria:

* Any teeth with microcracks or fracture lines
* Affected teeth without completed root canal treatment
* The defect was less than ¼ of crown or more than ¾ of the crown and the margin of the residual crown was more than 1 mm below the gingival level
* Poor oral hygiene and periodontal status which persisted or worsened after periodontal therapy and education
* Bruxism or clenching patients
* Poor general health or pregnancy
* Patients who have read the informed consent form and refused to be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of two materials | 36 months
  36 months-Modified United States Public Health Service

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided